CLINICAL TRIAL: NCT04162236
Title: Cardiac Dysfunction and Remodeling in Patients With Preeclampsia Regulated by Antiangiogenic Environment: Clinical and Experimental Approach
Brief Title: Cardiac Dysfunction and Remodeling in Patients With Preeclampsia
Acronym: ANGIOCOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-PRE-2019-63
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Preeclampsia; Cardiovascular Risk Factor; Pregnancy Complications
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications | interventions — Hematologic Tests; Carotid Intima-Media Thickness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, Placental samples, umbilical cord samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High Risk of Preeclampsia: Women with a singleton pregnancies attending for prenatal care in the maternal and fetal Medicine Unit will be asked to participate if they meet the following criteria:
  1)High risk for preeclampsia according to first trimester screening (maternal risk factors, blood preassure, PPAP-A, mean pulsatility index (PIm) of the uterine arteries (UtA) at 11.0 to 13.6 weeks of gestation (n=280).
  Women in this group will be subdivided in cases and controls according to the later development of preeclampsia:
  * cases: women developing PE (estimated n=40)
  * controls: women not developing PE (estimated n=240)
  Interventions: Diagnostic Test: Ecocardiographyc ultrasound
- Patients with Preeclampsia: Women with a singleton pregnancies attending for prenatal care in the maternal and fetal Medicine Unit will be asked to participate if they develop PE. Inclusion criteria: Patients presented with clinical signs and symptoms of preeclampsia (N=60).
  Interventions: Diagnostic Test: Ecocardiographyc ultrasound
- Control group: Healthy pregnant women with at low risk PE screening at 11.0 to 13.6 weeks of gestation (n=100).
  Interventions: Diagnostic Test: Ecocardiographyc ultrasound

INTERVENTIONS:
Diagnostic Test: Ecocardiographyc ultrasound — * Epidemiological data: Maternal history risk factors. First trimester scan is performed on all patients.
  * Antropomethric measures
  * Systemic arterial stiffness: using applanation tonometry with pulse wave analysis and pulse wave velocity.
  * Carotid Intima Thickness
  * Echocardiography assessment: It will be performed by a cardiologist specialized in cardiac imaging according to the usual standard protocol. High resolution images will be acquired and post-processed with dedicated software for the speckle tracking analysis. 2D echocardiography parameters to be acquired, tissue Doppler and speckle tracking software
  * Markers in maternal blood: Angiogenic factor and cardiac function biomarkers: Blood samples will be collected without anticoagulant to obtain serum. sFLT-1, PlGF, High-sensitivity Troponin and NT-proBNP will be measured using automated electrochemiluminescence immunoassays.
  Other Names: Blood test; Carotid intima thickness

SUMMARY:
Preeclampsia (PE) is a pregnancy-related hypertensive disorder drive by an anti-angiogenic environment. Women with PE have 2-4 time higher risk of developing cardiovascular disease (CVD), although the specific mechanism relating these two conditions remains elusive. In non-pregnant patients with coronary disease, angiogenic profile proved to be an independent predictor of poor prognosis and is associated with a higher mortality rate. The investigators hypothesized that in PE, the antiangiogenic environment determines the degree of cardiac dysfunction and remodeling and the posterior cardiovascular risk.

DETAILED DESCRIPTION:
Main objective: To determinie the relationship between antiangiogenic environment and cardioc dysfuntion and remodelin in women at risk and in established PE. M&M: placental dysfunction markers (angiogenic factors (PlGF) and anti-angiogenic factor (sFlt1) and cardiovascular risk variables (BMI, BP, arterial stiffness, copectin, proBNP, high-sensitivity troponin, carotid intima thickness and echocardiography parameters) would be evaluated in 280 patients at risk of PE according to first trimester screening and 100 controls. Additionally, cardiac dysfunction parameters would be evaluated in women with established PE (n=60) and common transcriptomic signatures between cardiovascular disease and preeclampsia would be investigated in placental samples from 10 PE and 10 controls. It will provide evidences to evaluate and characterize the association between angiogenic factors and cardiac dysfunction and remodeling in PE.

ELIGIBILITY:
Inclusion Criteria:

1. >18 and <45 years old.
2. Able to understand the study requirements.
3. Singleton pregnancy.
4. Accept of written informed consent.

Exclusion Criteria:

1. <18 or >45 years old.
2. Not able to understand the study requirements.
3. Multiple pregnancy.
4. Previous conditions: abnormal thrombophilia, alcohol or illicit drug use, type-1 diabetes, hyperthyroidism, renal disease, severe maternal illness, cytomegalovirus or toxoplasma infection, maternal HIV infection, , previous venous or arterial thrombotic event, and
5. known major fetal anomaly or chromosomal abnormality at inclusion
6. denial of written informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women at high risk of <preeclampsia on first trimestre scan
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
To prospectively assess both biochemical and biophysical markers of cardiovascular dysfunction in a cohort of patients with a risk of pe and in healthy pregnant women in the fisrt and third trimester of pregnancy. | 12 months
  - Cardiac dysfunction/remodeling in the first and third trimester of pregnancy and in 12 moths after delivery as defined by:
  1. abnormal cardiac performace in the ecocardiographyc ultrasound assessment or/and
  2. abnormal biochemical cardiac markers (copectin, proBNP, high-sensitivity troponin)

SECONDARY OUTCOMES:
To determine the correlation among antiogenic (PlGF) and anti-angiogenic factors (sFlt1) in maternal serum and biochemical and imaging markers of cardiac dysfunction and remodeling in patients with established PE AND | 9 months
  Venous blood will be drawn, with informed consent, from the cubital vein without a tourniquet and using a 20-G needle into Vacutainer CPT

OTHER OUTCOMES:
Determine cardiac dysfunction and metabolic status at 12 months after delivery and its correlation with cardiac and preeclampsia risk variables obtained during pregnancy | 12 months
To investigate angiogenesis and cardiovascular related genes in placental samples of women with preeclampsia and controls by microarrays and PCR validation. | 1 month
  Placenta will be collected at delivery time and tissue samples will be frozen in liquid N2 and fixed for histology and immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Llurba, Principal Investigator — Institut de Recerca Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ullmo J, Cruz-Lemini M, Bos-Real L, Padilla M, Coma-Barbara M, Martorell S, Mora J, Ordonez-Llanos J, Llurba E; AngioCor working group. Cardiovascular risk assessment in women at high risk for pre-eclampsia in first half of pregnancy. Ultrasound Obstet Gynecol. 2025 Jul;66(1):65-72. doi: 10.1002/uog.29247. Epub 2025 Jun 5. PMID 40471220
- [Derived] Ullmo J, Cruz-Lemini M, Sanchez-Garcia O, Bos-Real L, Fernandez De La Llama P, Calero F, Dominguez-Gallardo C, Garrido-Gimenez C, Trilla C, Carreras-Costa F, Sionis A, Mora J, Garcia-Osuna A, Ordonez-Llanos J, Llurba E. Cardiac dysfunction and remodeling regulated by anti-angiogenic environment in patients with preeclampsia: the ANGIOCOR prospective cohort study protocol. BMC Pregnancy Childbirth. 2021 Dec 8;21(1):816. doi: 10.1186/s12884-021-04263-w. PMID 34879854